CLINICAL TRIAL: NCT01192438
Title: A Pilot Study to Evaluate Magnetic Resonance Thermal Image-guided Laser-Induced Interstitial Thermal Therapy for Focal Ablation of Prostate Cancer
Brief Title: Laser Based Focal Ablation of Low Grade Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Visualase, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-364A
Record Dates: First submitted 2010-08-27; First posted 2010-09-01 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Low Grade Prostate Cancer
Keywords: prostate; cancer; ablation; laser-induced; focal therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Procedure/surgery (Experimental)
  Interventions: Procedure: Laser-based thermotherapy

INTERVENTIONS:
Procedure: Laser-based thermotherapy — MRI-guided transperineal placement of a laser probe into the prostate
  Other Names: Visualase, Inc

SUMMARY:
The purpose of this study is to evaluate the safety of MRI-guided laser-induced thermal therapy of biopsy confirmed low-risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male, 45 years of age or older
* Diagnosis of prostate adenocarcinoma
* Clinical stage T1c or T2a
* Gleason score of 7 or less
* A minimum of 12 biopsy cores sampled during diagnostic biopsy
* Three or fewer biopsy cores with prostate cancer
* No single biopsy core with greater than 50% of tumor involvement
* A radiographically visible prostate lesion on MRI with concordance to biopsy sextant
* A documented Karnofsky performance status of at least 70
* Estimated survival of 20 years or greater, as determined by treating physician
* Ability to give informed consent

Exclusion Criteria:

* Previous surgery, radiation, or androgen deprivation therapy for prostate cancer
* Presence of any condition (e.g., metal implant, shrapnel) not compatible with MRI
* History of previous pelvic radiation
* Severe lower urinary tract symptoms as measured by an International Prostate Symptom Score (IPSS) of 20 or greater. (See Appendix A)
* History of other primary non-skin malignancy within previous three years

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Within 6 months of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Eggener, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States